CLINICAL TRIAL: NCT04536974
Title: The "Self Evaluation of Food Intake" (SEFI) as a Screening Test for Hospital Malnutrition in Children Over 10 Years
Acronym: SEFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_3019_SEFI; 2020-A00739-30 (Other: French national agency for drugs)
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Malnutrition, Child
Keywords: MALNUTRITION; CHILDREN; SEFI
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SEFI tool — Detect the risk of malnutrition with the SEFI tool

SUMMARY:
The goal is to find a simple tool that can be used by medical and paramedical staff and that is reliable to identify children at risk for malnutrition.

DETAILED DESCRIPTION:
The Ingesta Easy Assessment Score (SEFI®) (formerly "food intake assessment tool or EPA®") is validated in hospitals in adults to detect the risk of malnutrition and guide nutritional management. SEFI® combines a visual analogue scale (VAS) with a visual assessment of the portions consumed (www.sefi-nutrition.com). It comes in the form of a ruler equipped with a cursor and allows a visual assessment, by the patient himself, of his food intake, using an analog scale, or a choice of portions. consumed (see appendix). A score <7/10 is associated with malnutrition or the risk of malnutrition.

The investigators hypothesize that, in pediatric services for children 10 years of age or older, SEFI® would be a feasible and reliable tool for screening for the risk of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 to 17 and hospitalized in pediatric or pediatric surgery, regardless of the reason for hospitalization.
* Whose holders of parental authority have received information on the protocol and have not expressed their opposition to the child's participation in the study,
* Having received information on the protocol and not having expressed opposition to participating in the study.

Exclusion Criteria:

* Patients whose level of understanding does not allow the use of SEFI®

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 10 to 17 and hospitalized in pediatric or pediatric surgery, regardless of the reason for hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 680 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-03-18 (Estimated); Study Completion 2024-06-18 (Estimated)

PRIMARY OUTCOMES:
Assess the reliability of SEFI® for detecting the risk of acute malnutrition in pediatrics | 6 month
  rate of agreement between the diagnoses of malnutrition obtained by the SEFI® tool and those obtained by diagnostic tools already validated in children: the Weight to Height ratio (or Waterlow index)

SECONDARY OUTCOMES:
reliability of SEFI ® to detect the risk of chronic undernutrition in pediatrics | 6 months
  rate of agreement between the diagnoses of malnutrition obtained by the SEFI® tool and those obtained by diagnostic tools already validated in children: Weight to Age ratio and Height to Age ratio
feasibility of SEFI® | 6 months
  Percentage of completion of the test compared to the number of subjects included in the study (if the test is carried out for each person included = 100% feasibility)
correlations of VAS results (score or portions consumed) with occurrence of complications and length of hospital stay | 9 months
  Duration of hospitalization and complications during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Gauthier Foulon, Doctor, Principal Investigator — Rennes University Hospital
Locations (5):
- France (5):
  - CHU Angers, Angers
  - APHP Trousseau Paris University Hospital, Paris
  - Rennes University Hospital, Rennes
  - CHU Toulouse, Toulouse
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: Undecided